CLINICAL TRIAL: NCT05778435
Title: The Effect Of The Wireless Fetal Monitoring Used During Birth On The Women's Comfort, Labour Pain And Birth Satisfaction
Brief Title: The Effect of Wireless Fetal Monitoring System on Comfort, Pain and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Demet Cakir, Assist.Prof.Dr., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TRTOKAT60
Record Dates: First submitted 2022-12-28; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy Related
Keywords: Pain; Birth; Chilbirth Satisfaction; Wireless Fetal Monitoring; Comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- wireless fetal monitoring group (Experimental): wireless fetal monitoring system was applied to the experimental group
  Interventions: Device: wireless fetal monitoring system
- Control group (No Intervention): Standard wired fetal monitoring system was applied to the control group.

INTERVENTIONS:
Device: wireless fetal monitoring system — The wireless fetal monitoring system shortens the period of labor by enabling the woman to be more mobile during the intrapartum period.
  Arms: wireless fetal monitoring group

SUMMARY:
Wireless EFM shortens labor duration, increases birth satisfaction, and reduces perceived pain during labor. With wireless EFM, comfort in labor increases and higher labor comfort increases birth satisfaction. As perceived pain in labor decreases, birth satisfaction increases. Therefore, wireless EFM practice is recommended during the antepartum and intrapartum periods.

DETAILED DESCRIPTION:
Problem Wired Electronic Fetal Monitoring (EFM) limits the woman's freedom of movement during labor, causes inability to cope with labor pain, lack of comfort, and a decrease in labor satisfaction.

Background While EFM is performed as wired and wireless in the antepartum and intrapartum periods, wired application is common in the world and in our country.

Aim This randomized controlled study was conducted to evaluate the effect of the wireless fetal monitoring, which is used during birth, on the woman's comfort, labor pain and birth satisfaction.

Methods The study population consisted of 88 women, divided into two groups the experimental group (n=44) and the control group (n=44). The data were collected with the Personal Information Form, Childbirth Comfort Questionnaire (CCQ), Visual Pain Scale (VAS), and Birth Satisfaction Scale-Revised (BSS-R). During the intrapartum period, the wireless fetal monitoring system was used in the experimental group and the wired fetal monitoring system was used in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are willing to participate in the study,
* Aged 18-40 years,
* Having a healthy pregnancy,
* With a gestational age of > 37+0 weeks,
* With a cervical dilatation of 4-5 cm,
* With a singleton pregnancy,
* With a live fetus,
* Can speak Turkish,
* Do not have comprehension, perception, and communication problems participated in the study.

Exclusion Criteria:

* Pregnant women who did not comply with the study had communication problems,
* Had complications,
* Needed urgent cesarean delivery and wanted to withdraw from the study were excluded from the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Childbirth Comfort Questionnaire | When the cervical dilatation of the pregnant woman was 8-10 cm in labor, the CCQ were filled out by the researcher between contractions, when the pregnant feels good.
  The participants rated the questionnaire through a Likert-type scale ranging from 1 to 5. The scores that can be obtained from the scale vary from 9 to 45. Higher scores indicate higher comfort during labor, whereas lower scores mean lower comfort
Visual Analogue Scale | When the cervical dilatation of the pregnant woman was 8-10 cm in labor, the VAS were filled out by the researcher between contractions, when the pregnant feels good.
  To measure the level of the pain, mostly a 10-cm-long vertical or horizontal line labeled from "No pain" to "Unbearable pain" is used. The participants are asked to mark their pain level on the line by a line, dot, or simply showing. The distance between the "no pain" point and the marked point indicates the level of pain
Birth Satisfaction Scale-Revised | The BSS-R was conducted 1 h after the mother was taken from the labor room to the gynecology and obstetrics service. The time required for the rest need of the postpartum mother, to meet her personal needs and breastfeed her baby was also provided
  The lowest and the highest scores that can be obtained from the scale were 0 and 40, respectively. Higher scores indicate higher satisfaction. Satisfaction is classified as low satisfaction (0-13), medium satisfaction (14-27), and high satisfaction (28-40). The scale is implemented within the first three days after delivery birth.

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Dağlar, Principal Investigator — Cumhuriyet University; Demet Çakır, Principal Investigator — Cumhuriyet University
Locations (1):
- Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] van den Heuvel JFM, Teunis CJ, Franx A, Crombag NMTH, Bekker MN. Home-based telemonitoring versus hospital admission in high risk pregnancies: a qualitative study on women's experiences. BMC Pregnancy Childbirth. 2020 Feb 4;20(1):77. doi: 10.1186/s12884-020-2779-4. PMID 32019499
- [Background] Menihan CA, Kopel E. Electronic Fetal Monitoring: Concepts and Applications. 2nd Ed. Chapter 2. Philadelphia, Lippincott: Williams&Wilkins; 2008.
- [Background] Monson M, Heuser C, Einerson BD, Esplin I, Snow G, Varner M, Esplin MS. Evaluation of an external fetal electrocardiogram monitoring system: a randomized controlled trial. Am J Obstet Gynecol. 2020 Aug;223(2):244.e1-244.e12. doi: 10.1016/j.ajog.2020.02.012. Epub 2020 Feb 20. PMID 32087146
- [Background] Alfirevic Z, Stampalija T, Medley N. Fetal and umbilical Doppler ultrasound in normal pregnancy. Cochrane Database Syst Rev. 2015 Apr 15;2015(4):CD001450. doi: 10.1002/14651858.CD001450.pub4. PMID 25874722
- [Background] Mugyenyi GR, Atukunda EC, Ngonzi J, Boatin A, Wylie BJ, Haberer JE. Functionality and acceptability of a wireless fetal heart rate monitoring device in term pregnant women in rural Southwestern Uganda. BMC Pregnancy Childbirth. 2017 Jun 8;17(1):178. doi: 10.1186/s12884-017-1361-1. PMID 28595604
- [Background] van den Heuvel JFM, Ganzevoort W, De Haan-Jebbink JM, van der Ham DP, Deurloo KL, Seeber L, Franx A, Bekker MN. HOspital care versus TELemonitoring in high-risk pregnancy (HOTEL): study protocol for a multicentre non-inferiority randomised controlled trial. BMJ Open. 2019 Oct 28;9(10):e031700. doi: 10.1136/bmjopen-2019-031700. PMID 31662396
- [Background] Mhajna M, Schwartz N, Levit-Rosen L, Warsof S, Lipschuetz M, Jakobs M, Rychik J, Sohn C, Yagel S. Wireless, remote solution for home fetal and maternal heart rate monitoring. Am J Obstet Gynecol MFM. 2020 May;2(2):100101. doi: 10.1016/j.ajogmf.2020.100101. Epub 2020 Mar 17. PMID 33345967
- [Background] Rubarth LB, Schoening AM, Cosimano A, Sandhurst H. Women's experience of hospitalized bed rest during high-risk pregnancy. J Obstet Gynecol Neonatal Nurs. 2012 May-Jun;41(3):398-407. doi: 10.1111/j.1552-6909.2012.01349.x. Epub 2012 Apr 26. PMID 22537349
- [Background] Kent RA, Yazbek M, Heyns T, Coetzee I. The support needs of high-risk antenatal patients in prolonged hospitalisation. Midwifery. 2015 Jan;31(1):164-9. doi: 10.1016/j.midw.2014.08.003. Epub 2014 Aug 15. PMID 25193792
- [Background] Lawrence A, Lewis L, Hofmeyr GJ, Styles C. Maternal positions and mobility during first stage labour. Cochrane Database Syst Rev. 2013 Oct 9;2013(10):CD003934. doi: 10.1002/14651858.CD003934.pub4. PMID 24105444
- [Background] Nguyen K, Bamgbose E, Cox BP, Huang SP, Mierzwa A, Hutchins S, Caso B, Culjat M, Connelly C, Lacoursiere DY, Singh RS. Wearable Fetal Monitoring Solution for Improved Mobility During Labor & Delivery. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:4397-4400. doi: 10.1109/EMBC.2018.8513321. PMID 30441327
- [Background] Goncu Serhatlioglu S, Karahan N, Hollins Martin CJ, Martin CR. Construct and content validity of the Turkish Birth Satisfaction Scale - Revised (T-BSS-R). J Reprod Infant Psychol. 2018 Jul;36(3):235-245. doi: 10.1080/02646838.2018.1443322. Epub 2018 Mar 19. PMID 29553295
- [Background] Ryu D, Kim DH, Price JT, Lee JY, Chung HU, Allen E, Walter JR, Jeong H, Cao J, Kulikova E, Abu-Zayed H, Lee R, Martell KL, Zhang M, Kampmeier BR, Hill M, Lee J, Kim E, Park Y, Jang H, Arafa H, Liu C, Chisembele M, Vwalika B, Sindano N, Spelke MB, Paller AS, Premkumar A, Grobman WA, Stringer JSA, Rogers JA, Xu S. Comprehensive pregnancy monitoring with a network of wireless, soft, and flexible sensors in high- and low-resource health settings. Proc Natl Acad Sci U S A. 2021 May 18;118(20):e2100466118. doi: 10.1073/pnas.2100466118. PMID 33972445
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Alfirevic Z, Devane D, Gyte GM. Continuous cardiotocography (CTG) as a form of electronic fetal monitoring (EFM) for fetal assessment during labour. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD006066. doi: 10.1002/14651858.CD006066. PMID 16856111
- [Background] Delice K. Before Birth Of Pregnant, Memoır, Postpartum Evaluation Of Knowledge Level Of Satisfaction From Services (Elbistan Sample). Master's thesis, Beykent University, Social Sciences Institute, Department Of Business, Hospıtal And Health Institutions Management Department, Istanbul. 2019. https://tez.yok.gov.tr/UlusalTezMerkezi/tezDetay.jsp?id=1gk8TzmGFaXVQPYkrUU_4Q&no=Enb8wsxJlkjAQuCt4e2yfQ
- [Background] Coskuner Potur D, Dogan Merih Y. The Validity and Reliability of the Turkish Version of the Childbirth Comfort Questionnaire. Journal of Anatolia Nursing and Health Sciences. 2015;18(4):252-258.
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Martin CH, Fleming V. The birth satisfaction scale. Int J Health Care Qual Assur. 2011;24(2):124-35. doi: 10.1108/09526861111105086. PMID 21456488
- [Background] Roham M, Saldivar E, Raghavan S, Zurcher M, Mack J, Mehregany M. A mobile wearable wireless fetal heart monitoring system. In 2011 5th International Symposium on Medical Information and Communication Technology (pp. 135-138). IEEE. (2011, March).
- [Background] Akbas P, Ozkan Sat S, Is M, Yaman S. Turkısh Validity-Reliability Study Of The Scale Of For Coping With Labor Pain. Journal of Health Sciences of Kocaeli University. 2021;7(3):235-241.
- [Background] Pehlivan N, Demirel Bozkurt O. Vertıcal position in the second stage of labor: Vertical birth chair. Acta Medica Nicomedia. 2020;3(1):42-48.
- [Background] Schramm K, Lapert F, Nees J, Lempersz C, Oei SG, Haun MW, Maatouk I, Bruckner T, Sohn C, Schott S. Acceptance of a new non-invasive fetal monitoring system and attitude for telemedicine approaches in obstetrics: a case-control study. Arch Gynecol Obstet. 2018 Dec;298(6):1085-1093. doi: 10.1007/s00404-018-4918-y. Epub 2018 Sep 27. PMID 30264201
- [Background] WHO recommendations: Intrapartum care for a positive childbirth experience. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK513809/ PMID 30070803
- [Background] Essa MR, Hafez SK. Effect of different positions of pregnant women on their comfort and fetal cardiotocographic patterns during nonstress test. International Journal For Research in Health Sciences And Nursing. 2018;4(2):1-24.
- [Background] Watson K, Mills TA, Lavender T. Experiences and outcomes on the use of telemetry to monitor the fetal heart during labour: findings from a mixed methods study. Women Birth. 2022 May;35(3):e243-e252. doi: 10.1016/j.wombi.2021.06.004. Epub 2021 Jul 2. PMID 34219033
- [Background] Harkey KT, Casale MB, Pantelopoulos AA, Zurcher MA. Assessing the clinical use of a novel, mobile fetal monitoring device. Obstetrics & Gynecology. 2014;123:55S.
- [Result] Boatin AA, Wylie B, Goldfarb I, Azevedo R, Pittel E, Ng C, Haberer J. Wireless fetal heart rate monitoring in inpatient full-term pregnant women: testing functionality and acceptability. PLoS One. 2015 Jan 26;10(1):e0117043. doi: 10.1371/journal.pone.0117043. eCollection 2015. PMID 25622043
- [Result] Knupp RJ, Andrews WW, Tita ATN. The future of electronic fetal monitoring. Best Pract Res Clin Obstet Gynaecol. 2020 Aug;67:44-52. doi: 10.1016/j.bpobgyn.2020.02.004. Epub 2020 Mar 19. PMID 32299728